CLINICAL TRIAL: NCT00740649
Title: Single Ascending Dose Study Of The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of HSD-016 Administered Orally To Healthy Japanese Male Subjects
Brief Title: Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of HSD-016
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3248A1-1001
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — (R)-1,1,1-trifluoro-2-(3-((R)-4-(4-fluoro-2-(trifluoromethyl)phenyl)-2-methylpiperazin-1-ylsulfonyl)phenyl)propan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HSD-016
  Interventions: Drug: HSD-016
- 2 (Other): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HSD-016
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
This is a single ascending dose study of HSD-016 to provide the initial assessment of the safety, tolerability, how the drug is absorbed and eliminated, and it's effect on the body in Japanese male subjects.

ELIGIBILITY:
Inclusion:

1. Men, aged 20 to 45 years inclusive at screening.
2. Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight ≥45 kg
3. Healthy as determined by the investigator on the basis of screening evaluations.
4. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history.

Exclusion:

1. No presence or history of any disorder that may prevent the successful completion of the study.
2. No history of drug abuse within 1 year.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
clinical labs, adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Toshima-ku, Tokyo, Japan